CLINICAL TRIAL: NCT02146716
Title: Assessment of Energetic Resonance by Cutaneous Stimulation on Withdrawal Alcohol Symptoms.
Acronym: RESC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-840
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: RESC, alcohol withdrawal syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Energetic Resonance by Cutaneous Stimulation (Experimental): Energetic Resonance by Cutaneous Stimulation session in addition to standard treatment for patients with withdrawal alcohol symptoms.
  Interventions: Other: Energetic Resonance by Cutaneous Stimulation

INTERVENTIONS:
Other: Energetic Resonance by Cutaneous Stimulation — Energetic Resonance by Cutaneous Stimulation (RESC) is a non-invasive method based on energetic Chinese medicine principles and digital contact. RESC is characterized by echo phenomena between two stimulation points.
  Arms: Energetic Resonance by Cutaneous Stimulation

SUMMARY:
The purpose of RESC study is to assess the efficacy of Energetic Resonance by Cutaneous Stimulation on alcohol withdrawal symptoms measured by CUSHMAN score and in a second time to measure the benzodiazepine amount prescribed during the withdrawal time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 80 years,
* Patient with alcohol addiction,
* Patient needing alcohol withdrawal in a hospital.
* Patient with social Security,
* Patient with inform consent signed.

Exclusion Criteria:

* Pregnant women
* Minor.
* Major with guardianship.
* People without sufficient information because of troubles of cognitive functions, or without sufficient knowledge of French language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Cushman Score measure after Energetic Resonance by Cutaneous Stimulation | daily during one week
  CUSHMAN score is represented by a scale with 7 variables collecting physiological modifications or behavioural manifestations related to adrenergic answer, neurovegetative signs, confusion, nervousness, perceptive or hallucinatory phenomena.

SECONDARY OUTCOMES:
Anxiety depression scale | pre-screening, day 3 and day 7
prescribed benzodiazepine amount | day 0 to day 7
Analogic Visual Scale | before and after each Energetic Resonance by Cutaneous Stimulationsession at day 2, day 4 and day 6.
Quality of life scale | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Claude Augustin-Normand, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital croix rousse, Lyon, France